CLINICAL TRIAL: NCT02849262
Title: A Phase 2, Randomized, Vehicle-Controlled, Double-Blind, Parallel-Group Study to Explore the Pharmacodynamics, Safety and Efficacy of Topical Omiganan in Patients With External Genital Warts
Brief Title: Pharmacodynamics, Safety and Efficacy of Topical Omiganan in Patients With External Genital Warts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLS001-CO-PR-011
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Condylomata Acuminata (External)
MeSH Terms: conditions — Condylomata Acuminata | interventions — Omiganan; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omiganan (CLS001) (Experimental): CLS001 Topical Gel, 2.5%
  Interventions: Drug: Omiganan (CLS001) topical gel
- Vehicle (Placebo Comparator): Vehicle Topical Gel
  Interventions: Drug: Vehicle topical gel

INTERVENTIONS:
Drug: Omiganan (CLS001) topical gel
  Arms: Omiganan (CLS001)
Drug: Vehicle topical gel
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the pharmacodynamics, safety and efficacy of omiganan in patients with external genital warts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects ≥ 18 years of age, with external genital warts. The health status is verified by absence of evidence of any clinical significant active or uncontrolled chronic disease other than genital warts following a detailed medical history and a complete physical examination including vital signs and 12-lead ECG. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
2. Clinically diagnosed and biopsy confirmed external genital warts. Subject has at least 3 external genital warts.
3. Willing to give written informed consent and willing and able to comply with the study protocol.

Exclusion Criteria:

Eligible subjects must meet none of the following exclusion criteria at screening:

1. Clinically significant abnormalities, as judged by the Investigator, in laboratory test results including haematology, blood chemistry panel, virology or urinalysis. In the case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
2. Current clinically significant skin conditions in the anogenital area (e.g. atopic dermatitis, lichen sclerosus, lichen planus or psoriasis).
3. Pregnant, breast feeding or trying to conceive.
4. Participation in an investigational drug or device study within 3 months prior to screening or more than 4 times a year.
5. Loss or donation of blood over 500 mL within three months (males) or four months (females) prior to screening.
6. Use of active treatment (i.e. cryotherapy, laser therapy, topical medication and/or surgical treatments) for genital warts within 28 days prior to first study drug administration.
7. Immunosuppressed patients, having an immunodeficiency (primary or secondary, like HIV) or receiving immunosuppressive therapy (i.e. Transplant patients).
8. Males or Females who received a vaccination with Gardasil or Cervarix.
9. Any (medical) condition that would, in the opinion of the Investigator, potentially compromise the safety or compliance of the patient or may preclude the patient's successful completion of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Clinical Assessment (Visible Lesions) | 24 Weeks
  Count of all visible lesions
Clinical Assessment (Percent clearance of treated lesions) | 24 Weeks
Clinical Assessment (Reduction of wart size) | 24 Weeks
  Includes 2D and 3D photography
Clinical Assessment (PRO) | 24 Weeks
  Change in Patient-reported outcomes
Pharmacodynamics (Local Immunity Status) | 24 Weeks
  Histological changes
Pharmacodynamics (HPV Viral Load Assessment) | 24 Weeks
  Quantitative PCR including HPV genotyping in swabs, qPCR to assess change from baseline, mean HPV viral load at treatment weeks and overall

SECONDARY OUTCOMES:
Safety and Tolerability (e-diary) | 24 Weeks
  Compliance with dosing instructions (patient completed e-diary)
Safety (AE) | 24 Weeks
  Adverse Events will be collected throughout the study
Safety (Laboratory Safety Testing) | 24 Weeks
  Lab samples will be collected throughout the study
Safety (Treatment-emergent AE and SAE) | 24 Weeks
  Treatment-emergent AE and SAE will be collected throughout the study
Safety (Vital Signs) | 24 Weeks
  Vital Signs will be collected throughout the study
Safety (ECG) | Screening and End of Study
  ECGs will be collected at before beginning and end of study

CONTACTS AND LOCATIONS:
Locations (1):
- LUMC/Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rijsbergen M, Rijneveld R, Todd M, Feiss GL, Kouwenhoven STP, Quint KD, van Alewijk DCJG, de Koning MNC, Klaassen ES, Burggraaf J, Rissmann R, van Poelgeest MIE. Results of phase 2 trials exploring the safety and efficacy of omiganan in patients with human papillomavirus-induced genital lesions. Br J Clin Pharmacol. 2020 Nov;86(11):2133-2143. doi: 10.1111/bcp.14181. Epub 2020 Sep 28. PMID 31755993